CLINICAL TRIAL: NCT02470000
Title: Treatment of Chronic Myofascial Pain Syndrome Over Neck by Using Intravascular Laser Irradiation of Blood
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CMRPG8D0921
Record Dates: First submitted 2015-02-09; First posted 2015-06-12 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-07

CONDITIONS: Myofacial Pain Syndromes
Keywords: myofascial pain; neck; laser; elastography; shear wave velocity; randomized control trial; Intravascular Laser Irradiation of Blood
MeSH Terms: conditions — Facial Neuralgia | interventions — Transcutaneous Electric Nerve Stimulation; Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental Group (Experimental): Intravascular laser irradiation of blood (ILIB, output power 0.3mW), Transcutaneous electrical nerve stimulation (TENS), stretching exercise.
  Interventions: Device: Intravascular laser irradiation of blood (ILIB); Device: Transcutaneous electrical nerve stimulation; Other: Stretching exercise
- Control Group (Sham Comparator): Intravascular laser irradiation of blood (ILIB, output power 0mW), Transcutaneous electrical nerve stimulation (TENS), stretching exercise.
  Interventions: Device: Intravascular laser irradiation of blood (ILIB); Device: Transcutaneous electrical nerve stimulation; Other: Stretching exercise

INTERVENTIONS:
Device: Intravascular laser irradiation of blood (ILIB) — continuous-wave ILIB is performed using a 632.8nm (red light) laser beam from a He-Ne laser machine (Y-J ILIB-5, Bio Human Energy Cooperation, New Taipei City, Taiwan, R.O.C.).The participants sit on a sofa with their arms relax and supported on the table. A 24-gauge catheter is inserted to a superficial vein in upper extremity under sterile preparation, and an optic fiber channel is connected to the catheter for blood irradiation.
  Other Names: ILIB
Device: Transcutaneous electrical nerve stimulation — TENS over neck for 15 minutes.
  Other Names: TENS
Other: Stretching exercise — stretching exercise to the involved muscle for 15 minutes.

SUMMARY:
Myofascial pain syndrome (MPS) is characterized by single or multiple trigger points (TrP) in taut bands within the affected muscles. Chronic MPS over neck is prevalent and responsible for markedly loss of work-day and a reduction of quality of life.

Intravascular laser irradiation of blood (ILIB) involves in vivo illumination of the blood by low-level laser light through an optical fiber inserted in a vein. Researches disclosed that ILIB reduced blood viscosity, enhanced erythrocyte deformity, and increased oxygen saturation in blood. However, no research studies the effectiveness of ILIB to treat MPS.

Real-time sonoelastography (RTS) and shear wave velocity (SWV) are used to detect the stiffness of skeletal muscles. RTS is displayed as a color-coded graphic to represent the relative stiffness of structures. For a given material, faster SWV indicates the greater stiffness. To our knowledge, only one research using RTS and SWV to study MPS.

To elucidate the effectiveness of ILIB to treat chronic MPS over neck, and the validity of RTS and SWV for MPS, we conducted this study.

DETAILED DESCRIPTION:
1. Time interval of the study: from 2014-11-1 to 2016-10-31 2. Participants and sample size:

1. Participants: Patients having chronic MPS over neck were randomized allocated to experimental group or control group. Participants in both groups are evaluated before and after the interventions (week 0 and week 2 respectively), and 12 week after the intervention (week 14). Both participants and evaluators don't know the allocation.
2. Sample size: thirty-six participants. The investigators plan to recruit 18 participants in each year.

III. Intervention:

Participants in experimental group receive ILIB (He-Ne laser, wavelength 632.8nm) with output power 0.3mW for 60minutes and following transcutaneous electric nerve stimulation (TENS) and stretching exercise every day except weekend for 2 weeks. Participants in control group receive sham therapies with the same protocol but no laser energy output

IV.Outcome Measures:

1.Primary outcome: Pain as measured by using a 10-cm long visual analogue scale (0 indicates no pain while 10 indicates worst pain) at rest and at movement.

2.Secondary outcomes:

1. .Pressure pain threshold (PPT) as measured by a pressure algometer, Force Dial FDK 20 with a scale ranging from 0 to 10 kg (Wagner Instruments, Greenwich, USA). The participant is in sitting position and relaxes, and the most painful TrPs in the taut band is measured. The investigators follow the procedures of measurement described by Fischer. The PPT is defined as the minimal pressure that results in the sensation change from pressure to pain. The investigators perform 3 repetitive measurements at an interval of 20 seconds, and the mean values will be analyzed.
2. .Shear wave velocity (SWV): SWV is undertaken by a physiatrist specialized in musculoskeletal US using a US system with 4-9 MHz multifrequency linear transducer (S2000; Siemens Healthcare, Erlangen, Germany). The posture of participant is the same with which when testing PPT. The investigators minimize probe pressure on muscles to avoid affect muscle stiffness. SWV of bilateral upper trapezius (TPZ), levator scapulae (LS), sternocleidomastoid (SCM) and the most painful TrP in taut band are measured longitudinally while their B-mode image qualities are optimal. When measuring TPZ, the probe was located at the midpoint of occipital protuberance and acromion and the ROI was placed inside the muscle belly. The SWV of LS is measured at the midpoint of superior-medial border of scapulae and the C1 transverse process. For the measurement of SCM, the probe is positioned at the midpoint of sternum and mastoid process. The most painful TrP in taut band is recognized by the participants and then marked and recorded its position related to bony landmarks with a measuring tape. SWV of each muscle is measured 10 times, and the median of the 10 valid measurements will be analyzed.
3. .Real-time sonoelastography (RTS): RTS is accessed by the aforementioned physiatrist by using the US system. RTS is depicted on the right side of the screen, while the longitudinal 2D image on the most painful TrP in taut band is displayed on the left side. The compression force applied is adjusted according to a quality factor set on the machine, which is displayed on the screen. A quality factor ≧ 60 indicates optimal compression force. The investigator stores the representative image with a quality factor ≧ 60, and determines the RTS score. Later, the stored images are analyzed with ImageJ software (National Institutes of Health,Bethesda, USA). The area of taut band on image is selected, and color histograms are made and the means of the blue pixel and the red pixel are recorded. The color pixels range from 0 to 255. Intrarater and interrater reliability tests for RTS and SWV are undertaken in the first 10 participants.
4. . World Health Organization Quality of Life Questionnaire Short Form (WHOQOL - BREF) Taiwan Version: WHOQOL - BREF Taiwan Version consists of 4 domains (physical health, psychological, social relationship, and environment) and a total 28 items. Each item has a five-point Likert-type response scale, and four types of scale descriptors (capacity, frequency, intensity and evaluation) are used.37 Individual domain score and total QOL score can be calculated through straightforward summative scaling. A higher score indicates a better QOL. This questionnaire was proved to be reliable and valid for many diseases.

V. Analysis and Statistics: Reliability of RTS and SWV are tested by using intraclass correlation coefficients. Within-group and between-group comparisons are made by using a repeated-measure ANOVA. Correlation coefficients among outcomes are calculated.

ELIGIBILITY:
Inclusion Criteria:

* (1) age ≧ 18 years old; (2) willing to sign an inform consent; (3) having a chronic MPS over neck at least 6 months. The diagnosis of MPS was made while the following criteria are met: (a) recognized pain with exquisite spot tenderness on a palpable taut band over the pain area; (b) presence of one of the two confirmatory signs: referred pain and local twitch response

Exclusion Criteria:

* (1) pregnancy; (2) bleeding tendency; (3) active systemic infective or inflammatory disease; (4) major surgery or trauma in the recent 3 months; (5) unstable cervical spine; (6) rheumatoid arthritis34; (7) open wound over neck; (8) pace-maker or defibrillator implantation; (9) overt neuropathic pain or radiation pain; (10) inability to express pain or quality of life.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2014-11; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Pain | week 0, week 2, week 14
  Pain as measured by using a 10-cm long visual analogue scale (0 indicates no pain while 10 indicates worst pain) at rest and at movement.

SECONDARY OUTCOMES:
Pressure pain threshold (PPT) | week 0, week 2, week 14
  Pressure pain threshold (PPT) as measured by a pressure algometer, Force Dial FDK 20 with a scale ranging from 0 to 10 kg (Wagner Instruments, Greenwich, USA). The participant is in sitting position and relaxes, and the most painful TrPs in the taut band is measured. The investigators follow the procedures of measurement described by Fischer. The PPT is defined as the minimal pressure that results in the sensation change from pressure to pain. The investigators perform 3 repetitive measurements at an interval of 20 seconds, and the mean values will be analyzed.
Shear wave velocity (SWV) | week 0, week 2, week 14
  SWV is undertaken by using a US system with 4-9 MHz multifrequency linear transducer. The investigators minimize probe pressure on muscles to avoid affect muscle stiffness. SWV of bilateral upper trapezius (TPZ), levator scapulae (LS), sternocleidomastoid (SCM) and the most painful TrP in taut band are measured longitudinally while their B-mode image qualities are optimal. When measuring TPZ, the probe was located at the midpoint of occipital protuberance and acromion and the ROI was placed inside the muscle belly. The SWV of LS is measured at the midpoint of superior-medial border of scapulae and the C1 transverse process. For the measurement of SCM, the probe is positioned at the midpoint of sternum and mastoid process. The most painful TrP in taut band is recognized by the participants and then marked and recorded its position related to bony landmarks with a measuring tape. SWV of each muscle is measured 10 times, and the median of the 10 valid measurements will be analyzed.
Real-time sonoelastography (RTS) | week 0, week 2, week 14
  RTS is accessed by the aforementioned physiatrist by using the US system. RTS is depicted on the right side of the screen, while the longitudinal 2D image on the most painful TrP in taut band is displayed on the left side. The compression force applied is adjusted according to a quality factor set on the machine, which is displayed on the screen. A quality factor ≧ 60 indicates optimal compression force. The investigator stores the representative image with a quality factor ≧ 60, and determines the RTS score. Later, the stored images are analyzed with ImageJ software (National Institutes of Health,Bethesda, USA). The area of taut band on image is selected, and color histograms are made and the means of the blue pixel and the red pixel are recorded. The color pixels range from 0 to 255. Intrarater and interrater reliability tests for RTS and SWV are undertaken in the first 10 participants.
World Health Organization Quality of Life Questionnaire Short Form Taiwan Version: WHOQOL - BREF Taiwan Version | week 0, week 2, week 14
  WHOQOL - BREF Taiwan Version consists of 4 domains (physical health, psychological, social relationship, and environment) and a total 28 items. Each item has a five-point Likert-type response scale, and four types of scale descriptors (capacity, frequency, intensity and evaluation) are used.37 Individual domain score and total QOL score can be calculated through straightforward summative scaling. A higher score indicates a better QOL. This questionnaire was proved to be reliable and valid for many diseases.

CONTACTS AND LOCATIONS:
Overall Officials: Lin-Yi Wang, MD, Study Chair — Rehabilitation
Locations (1):
- Lin-Yi Wang, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Srbely JZ. New trends in the treatment and management of myofascial pain syndrome. Curr Pain Headache Rep. 2010 Oct;14(5):346-52. doi: 10.1007/s11916-010-0128-4. PMID 20607458
- [Background] Hoving JL, Gross AR, Gasner D, Kay T, Kennedy C, Hondras MA, Haines T, Bouter LM. A critical appraisal of review articles on the effectiveness of conservative treatment for neck pain. Spine (Phila Pa 1976). 2001 Jan 15;26(2):196-205. doi: 10.1097/00007632-200101150-00015. PMID 11154541
- [Background] Gur A, Sarac AJ, Cevik R, Altindag O, Sarac S. Efficacy of 904 nm gallium arsenide low level laser therapy in the management of chronic myofascial pain in the neck: a double-blind and randomize-controlled trial. Lasers Surg Med. 2004;35(3):229-35. doi: 10.1002/lsm.20082. PMID 15389743
- [Background] Bron C, Dommerholt JD. Etiology of myofascial trigger points. Curr Pain Headache Rep. 2012 Oct;16(5):439-44. doi: 10.1007/s11916-012-0289-4. PMID 22836591
- [Background] Yap EC. Myofascial pain--an overview. Ann Acad Med Singap. 2007 Jan;36(1):43-8. PMID 17285185
- [Background] Chung H, Dai T, Sharma SK, Huang YY, Carroll JD, Hamblin MR. The nuts and bolts of low-level laser (light) therapy. Ann Biomed Eng. 2012 Feb;40(2):516-33. doi: 10.1007/s10439-011-0454-7. Epub 2011 Nov 2. PMID 22045511
- [Background] Chow RT, Heller GZ, Barnsley L. The effect of 300 mW, 830 nm laser on chronic neck pain: a double-blind, randomized, placebo-controlled study. Pain. 2006 Sep;124(1-2):201-10. doi: 10.1016/j.pain.2006.05.018. Epub 2006 Jun 27. PMID 16806710
- [Background] Chow RT, Johnson MI, Lopes-Martins RA, Bjordal JM. Efficacy of low-level laser therapy in the management of neck pain: a systematic review and meta-analysis of randomised placebo or active-treatment controlled trials. Lancet. 2009 Dec 5;374(9705):1897-908. doi: 10.1016/S0140-6736(09)61522-1. Epub 2009 Nov 13. PMID 19913903
- [Background] Altan L, Bingol U, Aykac M, Yurtkuran M. Investigation of the effect of GaAs laser therapy on cervical myofascial pain syndrome. Rheumatol Int. 2005 Jan;25(1):23-7. doi: 10.1007/s00296-003-0396-y. Epub 2003 Dec 12. PMID 14673617
- [Background] Dundar U, Evcik D, Samli F, Pusak H, Kavuncu V. The effect of gallium arsenide aluminum laser therapy in the management of cervical myofascial pain syndrome: a double blind, placebo-controlled study. Clin Rheumatol. 2007 Jun;26(6):930-4. doi: 10.1007/s10067-006-0438-4. Epub 2006 Oct 5. PMID 17021664
- [Background] Huang SF, Tsai YA, Wu SB, Wei YH, Tsai PY, Chuang TY. Effects of intravascular laser irradiation of blood in mitochondria dysfunction and oxidative stress in adults with chronic spinal cord injury. Photomed Laser Surg. 2012 Oct;30(10):579-86. doi: 10.1089/pho.2012.3228. Epub 2012 Aug 14. PMID 22891782
- [Background] Wasik M, Gorska E, Modzelewska M, Nowicki K, Jakubczak B, Demkow U. The influence of low-power helium-neon laser irradiation on function of selected peripheral blood cells. J Physiol Pharmacol. 2007 Nov;58 Suppl 5(Pt 2):729-37. PMID 18204188
- [Background] Mi XQ, Chen JY, Zhou LW. Effect of low power laser irradiation on disconnecting the membrane-attached hemoglobin from erythrocyte membrane. J Photochem Photobiol B. 2006 May 1;83(2):146-50. doi: 10.1016/j.jphotobiol.2005.12.018. Epub 2006 Feb 14. PMID 16481193
- [Background] Mi XQ, Chen JY, Liang ZJ, Zhou LW. In vitro effects of helium-neon laser irradiation on human blood: blood viscosity and deformability of erythrocytes. Photomed Laser Surg. 2004 Dec;22(6):477-82. doi: 10.1089/pho.2004.22.477. PMID 15684746
- [Background] Kwon DR, Park GY, Lee SU, Chung I. Spastic cerebral palsy in children: dynamic sonoelastographic findings of medial gastrocnemius. Radiology. 2012 Jun;263(3):794-801. doi: 10.1148/radiol.12102478. Epub 2012 Apr 10. PMID 22495685
- [Background] Friedrich-Rust M, Romenski O, Meyer G, Dauth N, Holzer K, Grunwald F, Kriener S, Herrmann E, Zeuzem S, Bojunga J. Acoustic Radiation Force Impulse-Imaging for the evaluation of the thyroid gland: a limited patient feasibility study. Ultrasonics. 2012 Jan;52(1):69-74. doi: 10.1016/j.ultras.2011.06.012. Epub 2011 Jul 7. PMID 21788057
- [Background] Kang J, Kwon H, Cho J, Oh J, Nam K, Yoon S, Kang M, Lee S, Han S. Comparative study of shear wave velocities using acoustic radiation force impulse technology in hepatocellular carcinoma: the extent of radiofrequency ablation. Gut Liver. 2012 Jul;6(3):362-7. doi: 10.5009/gnl.2012.6.3.362. Epub 2012 May 2. PMID 22844566
- [Background] Maher RM, Hayes DM, Shinohara M. Quantification of dry needling and posture effects on myofascial trigger points using ultrasound shear-wave elastography. Arch Phys Med Rehabil. 2013 Nov;94(11):2146-50. doi: 10.1016/j.apmr.2013.04.021. Epub 2013 May 14. PMID 23684553
- [Background] Leong HT, Ng GY, Leung VY, Fu SN. Quantitative estimation of muscle shear elastic modulus of the upper trapezius with supersonic shear imaging during arm positioning. PLoS One. 2013 Jun 25;8(6):e67199. doi: 10.1371/journal.pone.0067199. Print 2013. PMID 23825641
- [Background] Bai M, Du L, Gu J, Li F, Jia X. Virtual touch tissue quantification using acoustic radiation force impulse technology: initial clinical experience with solid breast masses. J Ultrasound Med. 2012 Feb;31(2):289-94. doi: 10.7863/jum.2012.31.2.289. PMID 22298873
- [Background] Kuo WH, Jian DW, Wang TG, Wang YC. Neck muscle stiffness quantified by sonoelastography is correlated with body mass index and chronic neck pain symptoms. Ultrasound Med Biol. 2013 Aug;39(8):1356-61. doi: 10.1016/j.ultrasmedbio.2012.11.015. Epub 2013 May 15. PMID 23683408
- [Background] Nightingale K. Acoustic Radiation Force Impulse (ARFI) Imaging: a Review. Curr Med Imaging Rev. 2011 Nov 1;7(4):328-339. doi: 10.2174/157340511798038657. PMID 22545033
- [Background] Gerwin RD, Shannon S, Hong CZ, Hubbard D, Gevirtz R. Interrater reliability in myofascial trigger point examination. Pain. 1997 Jan;69(1-2):65-73. doi: 10.1016/s0304-3959(96)03248-4. PMID 9060014
- [Background] Zvereva KV, Grunina EA. [The negative effects of low-intensity laser therapy in rheumatoid arthritis]. Ter Arkh. 1996;68(5):22-4. Russian. PMID 9082591
- [Background] Yao G, Chung CW, Yu CF, Wang JD. Development and verification of validity and reliability of the WHOQOL-BREF Taiwan version. J Formos Med Assoc. 2002 May;101(5):342-51. PMID 12101852
- [Background] Lin MY, KP; Hwang, JS; Wang, JD. Scale descriptor selection for Taiwan-version of questionnaire of World Health Organization quality of life. Chinese J Public Health (Taipei). 1999;18:262-270.
- [Background] Hong CZ. Treatment of myofascial pain syndrome. Curr Pain Headache Rep. 2006 Oct;10(5):345-9. doi: 10.1007/s11916-006-0058-3. PMID 16945250
- [Background] Eby SF, Song P, Chen S, Chen Q, Greenleaf JF, An KN. Validation of shear wave elastography in skeletal muscle. J Biomech. 2013 Sep 27;46(14):2381-7. doi: 10.1016/j.jbiomech.2013.07.033. Epub 2013 Jul 30. PMID 23953670